CLINICAL TRIAL: NCT05108688
Title: Mirtazapine vs Sumatriptan in the Treatment of Postdural Puncture Headache Following Obstetric Surgery Under Spinal Anesthesia: A Randomized Controlled Trial
Brief Title: Mirtazapine vs Sumatriptan in the Treatment of Postdural Puncture Headache
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD 209/2021
Record Dates: First submitted 2021-10-21; First posted 2021-11-05 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Mirtazapine; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mirtazapine Therapy group (M group) (Active Comparator)
  Interventions: Drug: Mirtazapine
- Sumatriptan Therapy group (S group) (Active Comparator)
  Interventions: Drug: Sumatriptan
- Control group ( C group) (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Mirtazapine — Mirtazapine 30 mg tablet once daily for 3 successive days
  Arms: Mirtazapine Therapy group (M group)
Drug: Sumatriptan — Sumatriptan 50 mg tablet once daily for 3 successive days
  Arms: Sumatriptan Therapy group (S group)
Other: Placebo — Placebo tablets once daily for 3 successive days.
  Arms: Control group ( C group)

SUMMARY:
Postdural puncture headache (PDPH) is a potential complication after spinal anesthesia caused by traction on pain-sensitive structures from low cerebrospinal fluid pressure (intracranial hypotension) following a leak of cerebrospinal fluid at the puncture site. Symptoms of this condition include a bilateral frontal or occipital headache that is worse in the upright position, along with nausea, neck pain, dizziness, visual changes, tinnitus, hearing loss, or radicular symptoms in the arms.

This study will examine the efficacy of mirtazapine in in the treatment of PDPH after obstetric surgery under spinal anesthesia and compared its efficacy with that of sumatriptan.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II Patients.
* Patients undergoing obstetric surgeries under spinal anesthesia. and complaining from moderate-to-severe PDPH after 25G or 27G spinal needle puncture.

Exclusion Criteria:

* Refusal of the intervention or participation in the study.
* Patient under age of 18 years old.
* Psychiatric illness.
* Patients with a history of ischemic heart disease, pregnancy-induced hypertension, chronic hypertension, cardiac, vascular, liver or renal impairment.
* Patients with a history of migraine.
* Patients with known hypersensitivity to study drugs.
* Patients currently using ergotamine, monoamine oxidase inhibitors, or selective serotonin reuptake inhibitors.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of refractory headache ((number of patients)(n),% of patients) (refractory: failed intervention and conservative treatment) after 72 hours | 72 hours after intervention (Day 0)
  Incidence of refractory headache ((number of patients)(n),% of patients) (refractory: failed intervention and conservative treatment) after 72 hours after intervention (Day 0)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt